CLINICAL TRIAL: NCT00764543
Title: Ambulatory Blood Pressure Measurement in Children With Congenital Urine Flow Obstruction
Status: No longer available | Type: Expanded Access
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Department of Urology (Unknown)
Responsible Party: Principal Investigator, Nancy Rollins, Assoc Dean, University of Texas Southwestern Medical Center
Other Study IDs: 052005-008
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hydronephrosis; Multicystic-dysplastic Kidney
Keywords: Unilateral hydronephrosis; Multicystic-dysplastic Kidney
MeSH Terms: conditions — Hydronephrosis; Multicystic Dysplastic Kidney

INTERVENTIONS:
Device: 24-hour ambulatory blood pressure monitor — Patients will go home with the 24-hour ambulatory blood pressure monitor to be returned at the clinic after 24 hours.

SUMMARY:
PURPOSE - HYPOTHESIS:

Children with unilateral congenital urine flow impairment, who require surgery, have abnormal 24-hour ambulatory blood pressure measurements.

OBJECTIVES:

To Measure 24-hour ambulatory blood pressure in children who have unilateral hydronephrosis or multicystic-dysplastic kidneys.

To compare these blood pressure measurements between the children who require surgical correction and those who do not need surgical correction.

BACKGROUND:

With the introduction of ultrasound examinations of pregnant women, previously undetected abnormalities in the fetus are being detected. Dilatation of the kidney caused by congenital unilateral impairment to the urine flow either partial, presenting as unilateral hydronephrosis or complete, as seen in children with multicystic-dysplastic kidneys, id a common finding affecting approximately 1: 1,500 pregnancies (Cendron et al 1994). The majority of infants do not require surgery, with only 25% needing surgery by 18 months of age (Ransley 1991). However, i8n a few. There is an increase in renal dilatation which ultimately results in a reduction in renal function.

The decision to operate is dependent on changes in renal pelvic diameter observed on serial ultrasound scans and on renal function. This process is often lengthy an requ8ires numerous scans, which can be upsetting for parents and child. M<any techniques have been used to identify, early, those patients who will require surgery. These have included: Intra-0renal pressure measurements, renal function, and calyceal diameter (Feung L 1997). To date, none have shown to be better than ultrasound (Dhillion HK 1998).

Ambulatory blood pressure monitoring measures the blood pressure multiple times during a predefined period. It, therefore, more accurately reflects the continuous nature of blood pressure during both awake and sleep periods (Sorof JM 2001). Consequently, it may detect abnormalities in blood pressure that are missed on a single reading. This has been shown in the one previous study investigating ambulatory blood pressure and patient with multicystic dysplastic kidneys (Seeman T et al Eur J Pediatr 2001). In this study, 20% of the children studied had abnormal results when ambulatory blood pressure was monitored.

DETAILED DESCRIPTION:
Patients who have a unilateral congenital impairment to urine flow, either partially or complete, will be included in this study. Only patients of investigators will be recruited for this study. Patients will be identified during their first clinic visit to see the urologist. If determined to be an eligible study candidate, they will be invited to join the research study.

Children enrolled at three months of age will be seen on their 6th, 12th, and 24th month and will take home a 24-hour ambulatory blood pressure monitor on each visit.

Children enrolled at 6 to 18 months of age will be seen every six months until their 24th month. They will also take home a 24-hout blood pressure monitor on each visit.

When the patient is enrolled in the study, they will follow the study design outlined in TABLE 1. The Table outlines scheduled intervals of clinic visits during which clinic staff and physicians will provide the standard of care required by the child, radiology procedure(s) required by the child's condition, and the initiation of the research-specific procedure of 24-Hour Ambulatory Blood Pressure Monitoring. Each visit will take approximately 2-3 hours. All care outlined in TABLE 1 are the standard of care except for the 24-Hour Ambulatory Blood Pressure Monitoring.

Clinic visits will encompass vital sign measurements in w2hich a single Blood Pressure will be measured, physical exam by the physician, and physician/parent discussion abo9ut the child's medical condition. These selected activities are estimated to take 30-45 minutes.

The standard of care radiology procedures scheduled at regular intervals for children with urine out-flow obstruction include a Renal Ultrasound estimated to take 30 minutes and a MAG 3 Renogram (MAG3 is an acronym for mercapto acetyl tri glycine, a compound that is chelated with a radioactive element - technetium-99m) estimated to take 60 minutes.

The renal ultrasound will be scheduled every clinic visit. A renal ultrasound is an imaging method in which high frequency sound wave echoes are picked up and displayed on a Television Monitor. Radiology personnel can visualize the size, shape and position, as well as the blood flow and urine flow through the kidneys, ureters and bladder.

A MAG-3 renogram will be scheduled during the clinic visits when the child is 3, 12 And 24 months of age. A MAG-3 renogram is a scan used to measure kidney function. Pictures of the kidneys are taken with a special camera following a small injection of a radioactive material called TechneScan MAG3.

The 24-Hour Ambulatory Blood Pressure Monitoring will be scheduled at every clinic visit. This procedure is a RESEARCH PURPOSES only. The device used to monitor blood pressure is FDA-approved and will measure the blood pressure at regular intervals over a 24-hour period. Monitoring intervals during the day-time are every 20 minutes (6:00 a.m. - 10:59 p.m.) and night-time intervals are every one-hour (11:00 p.m. - 5:59 a.m.). This procedure entails several steps for the parent as outlined in Table 1. The monitoring results will be downloaded into a computer and will require professional interpretation by Dr.

Mouin Seikaly. The interpretation of results will include consideration of what is written in the 24-hour blood pressure diary.

The 24-Hour Ambulatory Blood Pressure Monitoring encompasses several steps (outlined in Table 1.) The estimated total time for the patient to have this procedure is approximately 55 minutes broken down into the following components: Setting up the monitor and fitting the child with the appropriate cuff - 20 minutes; parental instruction for operating and caring for the monitor at home - 20-30 minutes initially followed by 15 minutes at subsequent visits, return of the monitor - 20 minutes. It should be noted that the 24-Hour Ambulatory Blood Pressure Monitor will accompany the patient at each visit. Management time at home includes the time to maintain a diary of recorded activities, events and medication administration times while the child is being monitored. Although this time will vary for each child, we estimate that it will average about 30 minutes of time over the 24-hour period.

24-hour ambulatory blood pressure monitoring will be read and interpreted by Dr. Mouin Seikaly, a pediatric nephrologist at Children's Medical Center of Dallas. The urologist responsible for discussing care and leading care decisions will be blinded to the interpretive results of the24-Hour Blood Pressure Monitoring. Only after the study will this information be available. We plan to finish the study in five years. TABLE 2 provides information about age based "normal" blood pressure readings for children in the 50th percentile on the growth chart of each age group.

Subjects will exit the study when clinic visit and study activities at age 24 months are completed, or when they have undergone surgery to correct the out-flow obstruction, or if the child is withdrawn prematurely by the parent or study doctor.

Indications for surgery include:

1. An increase of renal pelvic diameter (in the anterior posterior diameter) on two consecutive scans.
2. A drop in renal function of more than 5%.
3. An abnormal blood pressure reading on the single clinic blood pressure observation.

Reasons for premature withdrawal from the study include:

1. Parent does not comply with keeping clinic appointments.
2. Parent does not comply with or is unable to comply with physician instructions for medication management and/or other healthcare activity needed for child.
3. Parent is unable to manage the 24 hour blood pressure monitor device at home.
4. Child is unable to tolerate the blood pressure monitoring despite numerous distraction, diversion and comforting activities.
5. A different treatment approach is warranted and deemed to be more advantageous for the child.
6. Parental decision to withdraw child from the study prior to completion of study activities.
7. The physician determines that it is unsafe for the child to continue in the study.
8. The child's medical condition changes so that it is no longer appropriate for the child to continue in this study.

ELIGIBILITY:
Inclusion Criteria:

* Children of all races and both sexes including Spanish-speaking under 24 months of age with unilateral hydronephrosis greater than 10-mm in anterior posterior diameter; multicystic-dysplastic kidney on ultrasound examination.

Exclusion Criteria:

* Children over 24 months of age who have undergone surgery and whose parents do not wish to be involved in the study.

Max Age: 24 Months | Sex: All
Age Groups: Child